CLINICAL TRIAL: NCT04991207
Title: An Open-label, Three Period, Fixed Sequence Study to Assess the Effect of a Single Dose of BIA 5 1058 400 mg on the Steady State Pharmacokinetics of Bosentan in Healthy Subjects Under Fasting Conditions
Brief Title: Effect of BIA 5-1058 400 mg on the Steady State Pharmacokinetics of Bosentan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-107; 2015-004350-17 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIA 5-1058 (Experimental): Treatment Period 1: Subjects were admitted to the clinical unit on Day 1. Subjects received a single oral dose of BIA 5 1058 400 mg (4 x 100 mg tablets) on Day 1 after an overnight fast of at least 8 hours. Subjects were discharged from the clinical unit on Day 4 (approximately 72 hours after dosing) barring any medical reasons for an extended clinical stay.
  Interventions: Drug: BIA 5-1058
- Bosentan (Active Comparator): Treatment Period 2: Subjects were admitted to the clinical unit on Day 1. Subjects received multiple (twice daily [b.i.d.]) oral doses of bosentan (Tracleer® 1 x 125 mg film coated tablet) approximately 30 minutes before each meal (breakfast and dinner) from Days 1 to 5. On Day 6 after an overnight fast of at least 8 hours, subjects received a single morning dose of bosentan (Tracleer® 1 x 125 mg film coated tablet). Subjects were discharged from the clinical unit on Day 9 (approximately 72 hours after last dosing) barring any medical reasons for an extended clinical stay.
  Interventions: Drug: bosentan
- BIA 5-1058 and Bosentan (Experimental): Treatment Period 3: Subjects were admitted to the clinical unit on Day 1. Subjects received multiple b.i.d. oral doses of bosentan (Tracleer® 1 x 125 mg film coated tablet) approximately 30 minutes before each meal (breakfast and dinner) from Days 1 to 5. On Day 6 after an overnight fast of at least 8 hours, subjects received a single concomitant dose of BIA 5 1058 400 mg (4 x 100 mg tablets) and bosentan (Tracleer® 1 x 125 mg film coated tablet). Subjects were discharged from the clinical unit on Day 9 (approximately 72 hours after last dosing) barring any medical reasons for an extended clinical stay.
  Interventions: Drug: BIA 5-1058; Drug: bosentan

INTERVENTIONS:
Drug: BIA 5-1058 — Oral BIA 5-1058 (Zamicastat) 100 mg tablets
  Other Names: Zamicastat
  Arms: BIA 5-1058; BIA 5-1058 and Bosentan
Drug: bosentan — Oral Tracleer (bosentan) 125 mg film coated tablets
  Other Names: Tracleer
  Arms: BIA 5-1058 and Bosentan; Bosentan

SUMMARY:
the purpose of this study is:

* To assess the effect of BIA 5 1058 400 mg on the PK of bosentan.
* To assess the effect of bosentan on the PK of BIA 5 1058

DETAILED DESCRIPTION:
This study was an open label, three period, fixed sequence study in healthy male and female subjects performed at a single study center.

The study comprised:

* Screening during Days -28 to -2 (both inclusive).
* Three treatment periods separated by a washout period of at least 10 days.

Duration of Treatment:

The duration of participation for each subject was approximately 2 months and 3 weeks (including the screening period).

ELIGIBILITY:
Inclusion Criteria:

Subjects who met the following criteria were considered eligible to participate/continue in the study:

* Provided signed and dated informed consent before any study specific procedures were conducted.
* Male and female subjects aged 18 to 45 years (both inclusive) at the Screening Visit.
* Healthy as determined by the Principal Investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12 lead electrocardiogram (ECG). If a vital sign or ECG assessment was outside of the reference range at the Screening Visit or baseline, the assessment could have been repeated once as soon as possible and in any cases before enrollment to rule out any error.
* Non-smoker or ex-smoker for at least 3 months prior to the Screening Visit.
* Body mass index (BMI) between 18.5 and 29.9 kg/m2 (both inclusive) at the Screening Visit and on admission to each treatment period.
* Negative test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti HBc), immunoglobulin M (IgM) anti-HBc, hepatitis C virus antibody (anti HCV) and human immunodeficiency virus (HIV) (Types 1 and 2) antibodies at the Screening Visit.
* Negative screen for alcohol and drugs of abuse at the Screening Visit and on admission to each treatment period.
* Subject had to be willing and able to be confined to the clinical unit and had to adhere to the study and lifestyle restrictions.
* Male subjects had to use together with his female partner/spouse a highly effective contraception form of birth control in combination with a barrier method throughout the clinical study period. And agreed not to father a child or to donate sperm starting at the Screening Visit and throughout the clinical study.
* Female subjects had to either be of non childbearing potential or had to use highly effective methods of contraception from at least 3 months before the Screening Visit and throughout the clinical study in combination with a barrier method.

Exclusion Criteria:

1. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue disease or disorders within 5 years before the first IMP administration.
2. Documented coronary artery disease (any of prior myocardial infarction, positive stress test, positive nuclear perfusion study, prior coronary artery bypass graft [CABG] surgery or percutaneous coronary intervention, angiogram showing at least 75% stenosis in a major coronary artery), acute coronary syndrome or current symptoms of myocardial ischemia and angina.
3. Clinically relevant surgical history involving the stomach and/or intestinal system, potentially affecting absorption of IMPs.
4. Any clinically relevant findings in the laboratory tests, particularly any abnormality in the coagulation tests or the liver function tests, as judged by the Principal Investigator, at the Screening Visit and on admission to each treatment period. If a laboratory assessment was outside of the reference range at the local laboratory at the Screening Visit or baseline, the assessment could have been repeated once as soon as possible and in any cases before enrollment to rule out laboratory error.
5. Subjects with alanine aminotransferase (ALT) > 1.0 x the upper limit of normal (ULN) and/or aspartate aminotransferase (AST) > 1.0 x ULN and/or total bilirubin > 1.0 x ULN (isolated bilirubin > 1.0 x ULN and 1.5 x ULN was acceptable if bilirubin was fractionated and direct bilirubin < 35%), as confirmed by subsequent repeat assessment, at the Screening Visit and on admission to each treatment period.
6. History of relevant atopy or drug hypersensitivity.
7. History of alcoholism or drug abuse.
8. History of drinking > 24 g (males) and > 12 g (females) of pure alcohol per day (10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months before first admission to the clinical unit.
9. Use of alcohol within 72 hours before the Screening Visit and from 48 hours before dosing until completion of the Follow-up Visit.
10. Significant infection or known inflammatory process at the Screening Visit or upon admission to all treatment periods, as judged by the Principal Investigator.
11. Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of the Screening Visit or upon admission to all treatment periods.
12. Subjects with blood pressure (BP) measurements (mean of triplicate) outside the ranges, at the Screening Visit or admission to the first treatment period:

    * Systolic BP (SBP) < 100 mmHg or > 140 mmHg
    * Diastolic BP (DBP) < 60 mmHg or > 90 mmHg
13. Symptomatic orthostatic hypotension (drop of > 20 mmHg in SBP and/or > 10 mmHg in DBP when moving from supine to standing position), together with other symptoms, e.g., dizziness, at the Screening Visit or admission to the first treatment period.
14. Abnormal fundoscopy.
15. Electrocardiogram (mean of triplicate) with corrected QT interval using the Fridericia's formula (QTcF) > 450 ms at the Screening Visit or admission to the first treatment period.
16. Having an estimated glomerular filtration rate (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft Gault formula and normalized to an average surface area of 1.73m2.
17. Previous use of BIA 5 1058.
18. Use of any investigational drug or participation in any clinical study within 60 days or 5 half life times, whichever was longer, before first administration of IMP.
19. Having received IMP in more than 3 studies within 12 months before the Screening Visit.
20. Donated or received blood within 56 days before first administration of IMP.
21. Donated or received plasma within 30 days before first administration of IMP.
22. History of any significant bleeding within the last 56 days prior to first administration of IMP.
23. Vegetarians, vegans or other medical dietary restrictions.
24. Not able to communicate reliably with the Principal Investigator.
25. Unlikely to comply with the requirements of the study.
26. Use of over the counter (OTC) medications (including oral natural health products, vitamin and herbal supplements) within 7 days before the first IMP administration until the Follow up Visit.

    Use of prescription medications that could have affected the safety or other study assessments, in the Principal Investigator's opinion, within 14 days before the first IMP administration until the Follow-up Visit. By exception, acetaminophen/paracetamol 1000 mg/day was permitted.

    CYP2B6, CYP2C8, CYP2D6, CYP3A4 (BIA 5-1058 metabolism) and CYP2C9, CYP2C19, CYP3A4 (bosentan metabolism): Use of inhibitors taken within 7 days before the first IMP administration and inducers taken within 28 days before first IMP administration.
27. Any known allergy or contra-indication to any of the IMPs or their content.
28. The subject was an employee or the close relative of an employee of the Sponsor or the Contract Research Organization (CRO) involved in the clinical study.
29. Vulnerable subjects, e.g., subjects kept in detention, protected adults under guardianship, trusteeship and soldiers or subjects committed to an institution by governmental or juridical order.

    If female:
30. Pregnant or breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum observed concentration (for BIA 5-1058) | Up to 2 months and 3 weeks
  PK parameters were determined for BIA 5-1058 and its metabolites in plasma following single dose administration in Treatment Period 1 and Treatment Period 3.
  Samples for PK assessments of BIA 5 1058, and metabolites were collected at pre-dose (Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)
Tmax - Time corresponding to occurrence of Cmax (for BIA 5-1058) | Up to 2 months and 3 weeks
  PK parameters were determined for BIA 5-1058 and its metabolites in plasma following single dose administration in Treatment Period 1 and Treatment Period 3. Samples for PK assessments of BIA 5 1058, and metabolites were collected at pre-dose (Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)
T½ - Apparent terminal elimination half life (for BIA 5-1058) | Up to 2 months and 3 weeks
  PK parameters were determined for BIA 5-1058 and its metabolites in plasma following single dose administration in Treatment Period 1 and Treatment Period 3. Samples for PK assessments of BIA 5 1058, and metabolites were collected at pre-dose (Treatment Period 3, Day 6) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)
Cmax,ss - Maximum observed concentration at steady state (for bosentan) | Up to 2 months and 3 weeks
  PK parameters were determined for bosentan and metabolites in plasma following multiple dose administration in Treatment Period 2 and Treatment Period 3. Samples for PK assessments of bosentan and metabolites were collected at pre-last dose (Treatment Period 2, Day 6 and Treatment Period 3, Day 6) and post-last dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)
Tmax,ss - Time corresponding to occurrence of Cmax,ss at steady state (for bosentan) | Up to 2 months and 3 weeks
  PK parameters were determined for bosentan and metabolites in plasma following multiple dose administration in Treatment Period 2 and Treatment Period 3. Samples for PK assessments of bosentan and metabolites were collected at pre-last dose (Treatment Period 2, Day 6 and Treatment Period 3, Day 6) and post-last dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)
T½,ss - Apparent terminal elimination half-life at steady state (for bosentan) | Up to 2 months and 3 weeks
  PK parameters were determined for bosentan and metabolites in plasma following multiple dose administration in Treatment Period 2 and Treatment Period 3. Samples for PK assessments of bosentan and metabolites were collected at pre-last dose (Treatment Period 2, Day 6 and Treatment Period 3, Day 6) and post-last dose at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60 and 72 hours (15 samples)

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL International - Early Phase Clinical Unit - Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided